CLINICAL TRIAL: NCT02120066
Title: Submacular Hemorrhage Associated With Retinal Arterial Macro Aneurysm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor of Ophthalmology, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kyorineye015
Record Dates: First submitted 2014-04-15; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Submacular Hemorrhage; Ruptured Retinal Arterial Macro Aneurysms
Keywords: Submacular hemorrhage; Vitrectomy; tissue- plasminogen activator
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrectomy (Other)
  Interventions: Procedure: Vitrectomy for submacular hemorrhage; Drug: subretinal injection of tissue-plasminogen activator

INTERVENTIONS:
Procedure: Vitrectomy for submacular hemorrhage
Drug: subretinal injection of tissue-plasminogen activator

SUMMARY:
Evaluation of surgical outcome of vitrectomy with subretinal injection of recombinant tissue-plasminogen activator for submacular hemorrhage associated with retinal arterial macroanuerysms.

ELIGIBILITY:
Inclusion Criteria:

* The patients with sub macular hemorrhage associated with ruptured retinal arterial macro aneurysms

Exclusion Criteria:

* The eyes with preretinal or intraretinal hemorrhage at the fovea
* The patients with follow-up less than 3 months

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Displacement of sub macular hemorrhage | one year
  Anatomical recovery detected funduscopy and optical coherence tomography

SECONDARY OUTCOMES:
Visual acuity | one year
  Visual recovery after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan

REFERENCES:
- See also: Related Info — http://www.eye-center.org